CLINICAL TRIAL: NCT03860363
Title: Experiences With Automated Surgical Drainage in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Centese, Inc. (Industry)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: CRD-1129
Record Dates: First submitted 2019-02-27; First posted 2019-03-01 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Hemorrhage
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Treatment Group: Patients selected to participate.
  Interventions: Device: Blood drainage post cardiac surgery

INTERVENTIONS:
Device: Blood drainage post cardiac surgery — Blood drainage post cardiac surgery with Thoraguard Surgical Drainage System.

SUMMARY:
The purpose of this study is to evaluate the Thoraguard Surgical Drainage System in a real-world clinical environment. It is believed that this system will offer functional and clinical benefits over the current standard of care system for the removal of surgical fluids following cardiac surgery. Observations, experiences, and outcomes in a single hospital setting will be collected for the Thoraguard Surgical Drainage System.

DETAILED DESCRIPTION:
The Thoraguard System is intended for use for drainage of blood, fluids, and gases following cardiac and thoracic surgery. The system consists of an electronic control module, drainage kit (fluid collection canister and drainage line), and chest tube kit with novel chest tube. The system continuously monitors chest tube and drainage line patency, automatically clears the chest tube and drainage line from build-up, and provides digital readings of fluid output trends. Additionally, the system has patient safety alarms to notify clinical staff of an unexpected event associated with post-operative drainage. These functions offer significant improvements over current standard of care. Reliable post-operative drainage, reduced workload, and decreased variability in chest tube maintenance procedures have the potential to increase patient safety, reduce complications, and improve patient experience.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age ≥ 18)
* Patient undergoing non-emergent cardiac surgery
* Anticipated requirement for mediastinal chest tube drainage

Exclusion Criteria:

* Emergency surgery
* Re-do surgery
* Prior cardiac surgery
* Congenital cardiac disease or deformation
* Transplant surgery
* Ventricular Assist Device Surgery
* Suspected pulmonary air leak
* Atrial fibrillation
* In the opinion of the investigator the patient is unsuitable for the study for any other legitimate reason including incarceration, pre-existing medical or psychiatric condition, or interfering medications
* Known previous or concurrent enrollment in a clinical trial that, in the opinion of the investigator, might interfere with the objectives of this clinical trial
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-emergent cardiac surgery patients undergoing one of the following procedures: coronary artery bypass grafting, aortic valve repair or replacement, mitral valve repair or replacement, ascending aortic surgery, a combination of these procedures, or in conjunction with additional procedures such as left ventricular aneurysm repair.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Device User Experience Survey | At study completion - approximate 6 months.
  The Device User Experience Survey is an unvalidated, Sponsor-generated questionnaire aimed to increase the Sponsor's understanding of the usability of the Thoraguard Surgical Drainage System. The questionnaire asks approximately 15 questions (includes yes/no responses, rating scales, and fill-in-the-blank sections) and is to be completed by the treating clinicians at the completion of the study. A summary of all treating clinician responses will be generated at the completion of the study to summarize the overall user experience with the device.

CONTACTS AND LOCATIONS:
Overall Officials: Jack Boyd, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karimov JH, Gillinov AM, Schenck L, Cook M, Kosty Sweeney D, Boyle EM, Fukamachi K. Incidence of chest tube clogging after cardiac surgery: a single-centre prospective observational study. Eur J Cardiothorac Surg. 2013 Dec;44(6):1029-36. doi: 10.1093/ejcts/ezt140. Epub 2013 Mar 21. PMID 23520232
- [Background] Balzer F, von Heymann C, Boyle EM, Wernecke KD, Grubitzsch H, Sander M. Impact of retained blood requiring reintervention on outcomes after cardiac surgery. J Thorac Cardiovasc Surg. 2016 Aug;152(2):595-601.e4. doi: 10.1016/j.jtcvs.2016.03.086. Epub 2016 Apr 14. PMID 27210474
- [Background] Halm MA. To strip or not to strip? Physiological effects of chest tube manipulation. Am J Crit Care. 2007 Nov;16(6):609-12. No abstract available. PMID 17962505
- [Background] Mahmood K, Wahidi MM. Straightening out chest tubes: what size, what type, and when. Clin Chest Med. 2013 Mar;34(1):63-71. doi: 10.1016/j.ccm.2012.11.007. Epub 2013 Jan 17. PMID 23411057
- [Background] Shalli S, Saeed D, Fukamachi K, Gillinov AM, Cohn WE, Perrault LP, Boyle EM. Chest tube selection in cardiac and thoracic surgery: a survey of chest tube-related complications and their management. J Card Surg. 2009 Sep-Oct;24(5):503-9. doi: 10.1111/j.1540-8191.2009.00905.x. PMID 19740284